CLINICAL TRIAL: NCT06866340
Title: Evaluation of the Functionality and Perception of the Injured Limb in the Rehabilitation Process of Orthopedic Patients Undergoing Surgical Treatment for Traumatic Wrist Fracture
Brief Title: Evaluation of Limb Function and Perception in Rehabilitation After Traumatic Wrist Fracture Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: HES-SO Valais-Wallis (Other)
Responsible Party: Sponsor
Other Study IDs: POLSO24 (L3057)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fractures; Rehabilitation; Body Perception
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to assess the functional and perceptual alterations of the affected limb during rehabilitation in adult orthopedic patients who underwent surgical treatment for distal radius fractures. The main questions it aims to answer are:

What is the correlation between functional and perceptual alterations of the affected limb at the beginning and end of rehabilitation? How do these alterations influence rehabilitation duration and effectiveness?

Participants will:

Complete the patient questionnaires ((QuickDASH and ALPQ). Undergo handgrip strength tests and digital dynamometer tests to assess forearm muscle strength.

Have their range of motion evaluated by a physiotherapist during outpatient visits.

No additional diagnostic or instrumental examinations are required beyond routine clinical practice. The study will recruit 100 adult patients, last 24 months, and provide insights into the role of body perception in rehabilitation after wrist fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Patients who have undergone surgical treatment with a volar approach for a traumatic distal radius fracture at IRCCS Ospedale Galeazzi - Sant'Ambrogio.
* Willingness and ability to provide written informed consent.

Exclusion Criteria:

* Pre-existing neurological, psychiatric, or cognitive disorders that could affect motor function or body perception.
* Previous fractures of the same limb.
* Pregnancy or breastfeeding (self-reported).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult orthopedic patients undergoing rehabilitation after surgical treatment for a traumatic distal radius fracture. Participants will be recruited from the Hand Surgery Unit at IRCCS Ospedale Galeazzi - Sant'Ambrogio (Milan, Italy).
  Eligible patients must have undergone volar approach surgery for an isolated wrist fracture and will start a structured rehabilitation program following a 5-week immobilization period.
  Excluded from participation are individuals with neurological, psychiatric, or cognitive disorders, prior fractures in the same limb, or those who are pregnant or breastfeeding.
  A total of 100 participants will be consecutively enrolled to ensure a representative sample for statistical analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between functional and perceptual alterations at the beginning and end of rehabilitation | Measured at T1 (start of rehabilitation) and T2 (end of rehabilitation, 4-10 weeks later)
  The study will evaluate the relationship between functional parameters (grip strength, range of motion, QuickDASH score) and perceptual parameters (ALPQ score for body perception).

SECONDARY OUTCOMES:
Effect of functional and perceptual alterations on rehabilitation duration and effectiveness | Measured at T0 (before rehabilitation, after immobilization), T1 (start of rehabilitation), and T2 (end of rehabilitation, 4-10 weeks later)
  Examines how initial functional and perceptual impairments influence:
  Rehabilitation duration (measured in weeks and number of therapy sessions). Rehabilitation effectiveness (difference in QuickDASH, ALPQ, strength, and range of motion scores between T1 and T2).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided